CLINICAL TRIAL: NCT02175329
Title: A Randomized Clinical Trial of 3-unit Posterior Zirconia-ceramic Fixed Dental Prosthesis (FDPs) Veneered With Layered and Milled (CAD-on) Veneering Ceramics
Brief Title: Clinical Investigation on Zirconia-ceramic Three-unit Bridges With CAD-on Veneering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAD-On
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2017-03

CONDITIONS: Three-unit Posterior Bridges
Keywords: CAD/CAM, three-unit posterior bridges, zirconia framework

ARMS (2):
- CAD/CAM veneering (Experimental): CAD/CAM manufactured e.max CAD veneers on zirconia framework
  Interventions: Device: CAD/CAM Veneering
- manually layered (Active Comparator): Manually layered veneering on CAD/CAM fabricated zirconia bridge framework
  Interventions: Device: Manually layered veneering

INTERVENTIONS:
Device: CAD/CAM Veneering — CAD/CAM fabricated zirconia bridge framework is veneered with CAD/CAM fabricated lithium disilicate ceramic veneer
  Arms: CAD/CAM veneering
Device: Manually layered veneering
  Arms: manually layered

SUMMARY:
60 bridge frameworks are CAD/CAM manufactured from zirconia-ceramic; 30 bridges are veneered with CAD/CAM fabricated lithium disilicate ceramic, 30 bridges are manually layered. The goal is to compare clinical survival , biological or technical behaviour of the restorations.

DETAILED DESCRIPTION:
Randomized prospective controlled clinical study with three-unit posterior bridges made of zirconia-ceramic to compare veneering with manually layering or CAD/CAM fabricated lithium disilicate ceramic veneers. The hypothesis is that there is no difference in clinical survival of the restorations and no difference in biological or technical behaviour.

ELIGIBILITY:
Inclusion Criteria:

* single missing posterior tooth with two adjacent posterior teeth
* no acute conservative or paradontal treatment need except for the teeth to be treated in the study
* sufficient oral hygiene

Exclusion Criteria:

* known allergies to components
* bruxism
* missing antagonist tooth
* pregnancy or lactation
* missing written consent
* patients which are not expected to be compliant
* severe systemic diseases
* untreated carious lesions
* untreated parodontitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinical success | 2 years
  Clinical success is defined as more than 95% survival of the restoration after 2 years.

SECONDARY OUTCOMES:
Restoration quality | 1 week, 1 year, 2 years, 3 years, 4 years, 5 years
  Characterisation of the restorations according to United States Public Health Services (USPHS) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bindl, Dr.med.dent., Principal Investigator — Universität Zürich
Locations (1):
- Universität Zürich, Zentrum für Zahn-, Mund- und Kieferheilkunde, Zurich, Switzerland